CLINICAL TRIAL: NCT04580758
Title: Fractional CO2 Laser Combined With Platelet Rich Plasma Fluid Versus Gel Form in Treatment of Atrophic Acne Scars: A Randomized Clinical Trial
Brief Title: Fractional CO2 Laser Combined With PRP Fluid Versus Gel in Treatment of Acne Scars
Acronym: PRP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yasmine Ahmed Abd El-Maguid El-Hadidy (Other)
Responsible Party: Sponsor-Investigator, Yasmine Ahmed Abd El-Maguid El-Hadidy, Dermatology Resident, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kasr El Aini Hospital
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Atrophic Acne Scar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fractional laser with PRP fluid (Active Comparator): Fractional CO2 laser then the PRP is injected afterwards
  Interventions: Combination Product: Fractional laser with PRP fluid or PRP gel
- Fractional laser with PRP gel (Active Comparator): Fractional CO2 laser then the PRP gel is injected afterwards
  Interventions: Combination Product: Fractional laser with PRP fluid or PRP gel

INTERVENTIONS:
Combination Product: Fractional laser with PRP fluid or PRP gel — 20 participants divided into 2 groups of 10 10 participants will do Fractional laser with PRP fluid sessions and 10 participants will do Fractional laser with PRP gel

SUMMARY:
This study is to test the efficacy of fractional laser combined with either PRP fluid or PRP gel in the treatment of atrophic acne scars

DETAILED DESCRIPTION:
The study will include 20 patients, treated with fractional CO2 laser plus PRP fluid on one side of the face and fractional CO2 laser plus PRP gel on the other side.

Choosing which side of the face will be injected with PRP fluid and which side will be injected with PRP gel will be chosen according to a randomization table for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Both genders
* Skin types III - V
* Willingness and ability to comply with the requirements of the protocol
* Atrophic acne scars

Exclusion Criteria:

* Patients with active acne
* Patients with herpes labialis, bacterial infections, other infections such as HBV. HCV or HIV.
* Oral isotretinoin use in the previous 6 months
* Pregnancy
* Tendency to keloid formation
* Patients with severe systemic illness or malignancy
* Patients with connective tissue diseases
* Patients with bleeding tendencies or any other hematological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Test which combination is more effective, fractional laser with PRP fluid or fractional laser with PRP gel | one year
  Effectiveness of each combination will be measured with OCT, depth of a fixed scar on each side of the face will be measured at baseline and then compared with 1 month after the last session and 3 months after the last session

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided